CLINICAL TRIAL: NCT04824391
Title: Phase 2 Study for the Determination of Efficacy, Immunogenicity and Safety of Two Different Strengths of the Inactivated COVID-19 Vaccine ERUCOV-VAC, in a Placebo Controlled, Randomized, Double Blind Study Design.
Brief Title: Efficacy, Immunogenicity and Safety of Inactivated ERUCOV-VAC Compared With Placebo in COVID-19
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Health Institutes of Turkey (Other Government)
Collaborators: TC Erciyes University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: IDEAL00620-EU02-PK537-3
Record Dates: First submitted 2021-03-25; First posted 2021-04-01 (Actual); Last update posted 2023-08-03 (Actual); Status verified 2023-02

CONDITIONS: COVID-19
Keywords: COVID-19; Vaccine; Inactive; Phase 2
MeSH Terms: conditions — COVID-19; Sedentary Behavior | interventions — TURKOVAC; Vaccines

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- 3 mcg/0.5 ml Vaccine (Experimental): Low dose vaccine
  Interventions: Biological: ERUCOV-VAC 3 µg/0.5 ml Vaccine
- 6 mcg/0.5 ml Vaccine (Experimental): Medium dose vaccine
  Interventions: Biological: ERUCOV-VAC 6 µg/0.5 ml Vaccine
- Placebo (Placebo Comparator): Placebo
  Interventions: Other: Placebo

INTERVENTIONS:
Biological: ERUCOV-VAC 3 µg/0.5 ml Vaccine — Two IM applications on Days 1 and 28
  Arms: 3 mcg/0.5 ml Vaccine
Biological: ERUCOV-VAC 6 µg/0.5 ml Vaccine — Two IM applications on Days 1 and 28
  Arms: 6 mcg/0.5 ml Vaccine
Other: Placebo — Two IM applications on Days 1 and 28
  Arms: Placebo

SUMMARY:
The objective is to determine the efficacy, immunogenicity and safety of two different strengths (3 µg and 6 µg) of an inactivated COVID 19 Vaccine compared to placebo so that to demonstrate the efficacy and safety in prophylaxis of COVID-19. A 3rd application will be performed to approximately the half of the volunteers who were administered 3 μg/0.5 ml and who accept to be vaccinated for a 3rd time, on their month 4 visit.

ELIGIBILITY:
Inclusion Criteria:

* healthy Caucasian origin
* accepting not to participate in another COVID-19 vaccine study until the end of the study
* volunteers who do not plan to get a child in the next one year; the volunteer and the partner should use a reliable form of contraception (abstinence, condom, birth control implant, birth control pills used or IUD used by the partner) during the study for at least 1 year
* female participants of childbearing potential (defined as any female who has experienced menarche and who is NOT surgically sterile [ie, hysterectomy, bilateral tubal ligation, or bilateral oophorectomy] or postmenopausal [defined as amenorrhea at least 12 consecutive months) must agree to be heterosexually inactive through 12 months after the first vaccination OR agree to consistently use any of the described methods of contraception from through 12 months after the first vaccination.
* male subjects agree to refrain from sperm donation from the time of first vaccination until 3 months after last vaccination
* participants must refrain from blood or plasma donation from the time of first vaccination until 3 months after last vaccination
* the outcome of the following examinations should be clinically insignificant: medical and surgical history (hypo-, hypertension, allergy, other diseases, major surgery, micturition, defecation, sleep, illness within the last 4 weeks prior to the start of the trial);
* life style and habits (consumption of alcohol, nicotine, coffee, tea, coke, special diet, drug abuse) should be normal/acceptable
* body temperature, pulse rate, blood pressure and respiratory rate should be normal/acceptable.
* laboratory examination (blood/serum examination: sodium, potassium, calcium, total protein, albumin, glucose, creatinine, BUN, total bilirubin, AST, ALT, GGT, ALP, haemoglobin, haematocrit, erythrocytes, Ieukocytes, platelet count; HBsAg, HIV-Ab, HCV-Ab should be normal/acceptable.
* antiSARS CoV 2 total antibody (including COVID-19 IgG and/or IgM) negative in serum.
* body weight in relation to height and age accepted BMI range 18.5 and 32 kg/m2 - both inclusive

Exclusion Criteria:

* women with a positive blood (β-HCG) pregnancy test
* lactating women
* history of COVID-19 infection or showing COVID-19 infection symptoms
* having had contact to people with known COVID-19 infection in the last 14 days
* having fever (> 37.4oC in the last 24 hours), dry cough or feeling tired and having aches and pains, nasal congestion, runny nose, sore throat and diarrhea.
* positive real time RT-PCR COVID-19 test.
* leukemia or neoplasm in history.
* persons with autoimmune diseases
* allergic diathesis or any clinically significant allergic disease (i.e. asthma)
* any condition that might impair the immune response
* recent or current immunosuppressive medication
* any other vaccine application 30 days before the first dose
* presence or a history of clinically significant cardiovascular, renal, hepatic, pulmonary, metabolic, endocrine, haematological, gastrointestinal, neurological, psychiatric or other major diseases;
* disruption of platelets or other blood clotting disorders, which may cause contraindications to intramuscular administration
* clinically significant illness within 4 weeks before the start of the study. Especially any acute or chronic illness seizures.
* any regular intake or administration of any prescribed systemic or topical medication within 2 weeks prior to the start of the study; in the case of intake or administration of any prescribed systemic or topical medication within 4 weeks before the start of the study because of an insignificant illness, this should be stated in the CRF.
* intake or administration of OTC medication (including herbal remedies) which may have an effect on the study according to the investigator within 2 weeks prior to the start of the study
* volunteers who received antiviral drugs, immunoglobulins or blood transfusions or any other investigational drug within 4 weeks prior to the first study product administration
* concomitant intake or administration of any systemic or topical drugs (including herbal remedies) on the application days
* treatment with any investigational drug (i.e., drug not yet approved) in the last 4 weeks before beginning of the trial
* medication with drugs known to alter organs or systems such as barbiturates, phenothiazines, cimetidine, omeprazole etc. within the last 1 month (4 weeks)
* donation of blood or plasma more than 450 ml within the last 2 months (8 weeks) or any amount within the last month (4 weeks)
* supine blood pressure, after resting for 5 min, higher than 140/90 or lower than 100/60 mmHg
* supine pulse rate, after resting for 5 min, outside the range of 50 - 100 beats/min
* supine respiratory rate, after resting for 5 min, outside the range of 15 - 18 breathings / min
* laboratory values (appendix 5) outside normal range with clinical relevance at entry examination
* alcohol abuse i.e. regular use of more than 2 units of alcohol per day or a history of alcoholism or drug/chemical abuse (one unit of alcohol equals ½ l of beer, 200 ml wine or 50 ml of spirits) or recovered alcoholics
* caffeine abuse i.e. regular use of more than 750 mg/day caffeine
* alcoholic or methylxanthine-containing beverages or foods (coffee, tea, coke, chocolate) and fruit-juice from 24 hours prior to each application
* smoking of more than 10 cigarettes or equivalent per day, no smoking before application
* vegetarian or any special diet due to any reason
* knowledge to have any type of parenterally transmitted hepatitis or carrier of the HBsAg (HBsAg test positive)
* HIV-Ab test positive
* Test on anti-HCV antibodies positive
* legal incapacity and/or other circumstances rendering the subject unable to understand the nature, scope and possible consequences of the study
* evidence of an uncooperative attitude.

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Non-pregnant women
Enrollment: 250 (Actual)
Dates: Start 2021-02-10 (Actual); Primary Completion 2022-03-11 (Actual); Study Completion 2022-03-30 (Actual)

PRIMARY OUTCOMES:
Serum IgG antibody levels specific for the SARS-CoV- 2 rS protein antigen(s) | 12 months
Neutralizing antibodies from microneutralization assay | 12 months
Blood levels of cytokines: TNF-α, IFN-γ, IL-2, IL-4, IL-5 and IL-6 | 12 months

SECONDARY OUTCOMES:
Adverse events | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Zafer Sezer, Assoc.Prof., Study Director — Co-Investigator
Locations (1):
- Erciyes University, Kayseri, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Ozdarendeli A, Sezer Z, Pavel STI, Inal A, Yetiskin H, Kaplan B, Uygut MA, Bayram A, Mazicioglu M, Unuvar GK, Yuce ZT, Aydin G, Aslan AF, Kaya RK, Koc RC, Ates I, Kara A. Safety and immunogenicity of an inactivated whole virion SARS-CoV-2 vaccine, TURKOVAC, in healthy adults: Interim results from randomised, double-blind, placebo-controlled phase 1 and 2 trials. Vaccine. 2023 Jan 9;41(2):380-390. doi: 10.1016/j.vaccine.2022.10.093. Epub 2022 Nov 22. PMID 36460536
- See also: Paper — https://doi.org/10.1016/j.vaccine.2022.10.093